CLINICAL TRIAL: NCT04612686
Title: Physiological Phenotyping of Frailty Using Magnetic Resonance Imaging
Brief Title: Characterising Frailty Using Magnetic Resonance Imaging
Acronym: PHENOFRIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Medical Research Council (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20039
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Frailty; Frailty Syndrome; Frail Elderly Syndrome
Keywords: Phenotype; Magnetic resonance imaging; MRI; Phenotyping; Elderly; Frail; Frailty; Fried; Physiological; Physiology; Female; Heart; Brain; Muscle; Strength; Power output; Fatigability; Cognition; Older persons; Pre-frail; Non-frail
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frail: At screening participants will be classed as frail if their Electronic Frailty Index score is >0.24 and if their Clinical Frailty Scale score is 6. This will be confirmed following the Fried frailty phenotype assessment made during the first visit to the University laboratory. Participants exhibiting 3 or more frailty components (slowness, weakness, weight loss, exhaustion, low physical activity) will be classed as frail.
  All participants will receive the same assessment procedures.
- Pre-frail: At the point of screening, participants will be classed as pre-frail if their Electronic Frailty Index score is 0.13-0.24 and if their Clinical Frailty Scale score is 4-5. This will be confirmed following the Fried frailty phenotype assessment made during the first visit to the University laboratory. Participants exhibiting 1 or 2 frailty components (slowness, weakness, weight loss, exhaustion, low physical activity) will be classed as pre-frail.
  All participants will receive the same assessment procedures.
- Non-frail: At the point of screening, participants will be classed as non-frail if their Electronic Frailty Index score is 0-0.12 and if their Clinical Frailty Scale score is 1-2. This will be confirmed following the Fried frailty phenotype assessment made during the first visit to the University laboratory. Participants exhibiting no frailty components (slowness, weakness, weight loss, exhaustion, low physical activity) will be classed as non-frail.
  All participants will receive the same assessment procedures.

SUMMARY:
Ageing is associated with the development of various negative conditions, such as frailty. Defined as a decreased ability to combat negative stressors (e.g. injury and illness), frailty is highly prevalent in elderly adults and significantly increases an individual's risk of adverse events such as falls, illness and death. The underlying physical characteristics of frailty are currently incompletely understood, with many previous studies focusing on one tissue (e.g. the brain) in isolation. However, frailty is known to affect many tissues simultaneously, and to further our insight into the biological basis of frailty and how to treat it, we must determine how different organs are affected at the same time.

The study will look at the physical characteristics of non-frail and frail elderly females (aged 65 years and over), who are attending geriatric clinics across the Nottingham University Hospitals NHS Trust. We will aim to recruit 51 participants with this cohort broken down into non-frail (n=17), pre-frail (n=17) and frail (n=17) subgroups. Participants will be allocated to these groups based on their Electronic Frailty Index, Clinical Frailty Scale and Fried frailty phenotype scores. All participants will undergo basic muscle function tests (grip strength, leg strength and muscle activity) and questionnaires on their first visit to University of Nottingham laboratories. At a second visit, they will then undergo one Magnetic Resonance Imaging (MRI) scanning session, at the Sir Peter Mansfield Imaging Centre within the University, to gather information about the structure and function of their heart, brain and skeletal muscle. MRI scan protocols will take approximately 45-60 mins. Data gathered from MRI scanning will be compared across non-frail, pre-frail and frail groups to investigate differences across frailty states, with the aim of highlighting the defining physical characteristics of the frail state which may help to develop future treatment interventions to combat the condition.

We hypothesise that frail females will present with common physical characteristics, the clustering of which will be indicative of frailty severity. We also hypothesise that certain physical traits present in the frail will not be present in the non-frail.

DETAILED DESCRIPTION:
The study will recruit females aged over 65 years (n=51), from those attending hospital clinics for older people at both campuses of Nottingham University Hospitals National Health Service (NHS) Trust. A member of the clinical care team working within the clinic will identify potential participants who are 'frail', 'mildly frail/vulnerable' and 'non-frail' using the Clinical Frailty Scale (measured as part of routine care), and the electronic Frailty Index. Clinic staff will make the initial approach to patients about the study and if the individual is interested in taking part, clinic staff will inform the research team. A researcher will then approach the interested individual and provide a study information sheet outlining study procedures. Potential participants will then be given a week to consider participating in the research.

If individuals wish to participate, they will be invited to the David Greenfield Human Physiology laboratories at the Queen's Medical Centre. Here, researchers will explain the study again to volunteers and answer any questions that they may have. Volunteers will be asked to sign an informed consent document prior to any other study procedures being undertaken. Participants will initially have their height and body mass recorded and will complete questionnaires assessing their suitability to have magnetic resonance imaging (MRI) scans, their cognitive ability and independence across activities of daily living.

Each participant's frailty status will be confirmed via the Fried Frailty phenotype assessment which will include a timed 15ft (4.57m) walk, hand grip strength, and questionnaires (Center for Epidemiologic Studies Depression Scale, Minnesota Leisure Time Activity Questionnaire). Participants who do not exhibit any frailty components will be classed as non-frail, those showing one or two frailty components will be classified as pre-frail, and those presenting three or more components will be classed as frail. These measures of frailty severity will take approximately 30 minutes to complete.

Knee extensor strength and power measurements will then be made. They will involve participants being seated in a chair and supported within the measuring apparatus (a padded chair with back support at 90°) using straps (similar to a seat belt) which go across their hips and shoulders. The participant's ankle will be positioned against a lever arm of the equipment and again held in place by a padded support. The isometric strength assessment will involve the participant pushing against the lever arm with maximum effort whilst it is fixed and unable to move. A total of 3 contractions lasting ~2 seconds will be performed with a 1 min rest between each. Muscle power and fatigue will be assessed on the same machine but this time the lever arm will move at a fixed rate. Participants will be asked to extend their leg (as if kicking a ball) 10 times with the lever arm speed at a slow speed (60 degrees per second) and 10 at a faster speed (180 degrees per second). These tests of muscle power output have been administered routinely to elderly volunteers in the literature and our laboratory. However, if these tests are not tolerable for participants, we will terminate the test. Knee extensor measurements will take approximately 30 minutes to complete.

Measurements of thigh muscle motor unit recruitment and motor control (a measure of the electrical activity within the muscle) will then be taken. Measurements will involve placing adhesive non-invasive ECG pads on to the participant's thigh, and a small (24-gauge) needle inserted into the thigh muscle to a depth of ~0.5-2.5cm (depending on amount of subcutaneous fat present). Participants will then be asked to gently contract their thigh muscle (the limb will not be in motion) and the electrical activity of the muscle will be measured. In total, this measure will take approximately 40 minutes to complete. Once completed, the electrodes will be removed and the needle insertion site covered with a small adhesive dressing. Muscle activity measures will take approximately 40 minutes to complete.

On a separate day, following the visit to the physiology laboratories, participants will be invited to the Sir Peter Mansfield Imaging Centre at the University of Nottingham. Here, they will undergo MRI scanning to gather images of the heart, brain, skeletal muscle and fat content within the body. Participants will be made comfortable on the scan table using pillows and pads to support their back, neck and joints. They will be asked to lie as still as possible during the scan protocol and occasionally perform some short breath holds (necessary to acquire certain scans). In total, the time spent in the scanner will be approximately 60 minutes. However, lying still within the MRI scanner for ~60 minutes may be burdensome for elderly participants. Therefore, we will offer short comfort breaks after 15 minutes and 40 minutes of scanning, during which participants may leave the scan room to use the bathroom and consume refreshments if needed. This will not affect the scan procedure or image collection.

ELIGIBILITY:
Inclusion Criteria:

* Females aged over 65 years of age attending Nottingham University Hospitals NHS Trust 'falls and bone health' and general geriatric clinics;
* Able to provide informed consent;
* Once 17 participants have been recruited to any of the three study groups (non-frail, pre-frail, frail) the study will be restricted to people in the remaining groups only;
* Good understanding of written and spoken English.

Exclusion Criteria:

* Metal within the body which could be affected by MRI;
* Any other contraindications for MRI scan (e.g. brain aneurysm clips, permanent pacemaker);
* Over 190.5 cm in height
* Inability to lie on back within the MRI scanner
* Mobility limitations which would prevent the individual transferring onto equipment
* Unable to speak or understand English;
* In receipt of end of life care;
* Lacking the mental capacity to understand the requirements of study participation and provide consent.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — female sex
Study Population: Participants will be identified from hospital clinics for older people, many of whom will be frail. Participants will be female, aged over 65 years and outpatients attending these clinics.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | Baseline (During visit to University physiology laboratory)
  Hand grip strength measured by a handheld dynamometer

SECONDARY OUTCOMES:
Whole body skeletal muscle volume | Baseline (During visit to Sir Peter Mansfield Imaging Centre - University of Nottingham)
  The volume of individual and groups of skeletal muscles within the body. Assessed using MRI scanning sequences.
Volumes of individual muscles in the lower limbs | Baseline (During visit to Sir Peter Mansfield Imaging Centre - University of Nottingham)
  The volume of individual lower limb muscles (e.g. thigh, calf). Assessed using MRI scanning sequences.
White/grey matter volumes of the brain | Baseline (During visit to Sir Peter Mansfield Imaging Centre - University of Nottingham)
  Global and regional volumes of white/grey matter within the brain. Assessed using MRI scanning sequences.
Cerebral perfusion | Baseline (During visit to Sir Peter Mansfield Imaging Centre - University of Nottingham)
  Blood perfusion throughout the brain tissue will be assessed using MRI scanning sequences.
Motor unit size and recruitment in thigh muscle | Baseline (During visit to University physiology laboratory)
  The size and recruitment of motor units with muscles of the thigh will be assessed using intramuscular electromyography techniques.
Cardiac stroke volume, ejection fraction and aortic strain of the heart | Baseline (During visit to Sir Peter Mansfield Imaging Centre - University of Nottingham)
  Variables associated with heart structure and function will be assessed using MRI scanning sequences.
Knee extension strength | Baseline (During visit to University physiology laboratory)
  Strength of the quadriceps muscles will be assessed using a Cybex dynamometer, during isometric contractions.
Walking speed | Baseline (During visit to University physiology laboratory)
  Walking speed will be assessed during a timed 15 ft (4.57 m) walk, as part of the Fried frailty phenotype assessment.
Clinical Frailty Scale | Initial patient screening (within clinic of Nottingham University Hospitals)
  The Clinical Frailty Scale will provide information on patient's frailty status already evident in their medical records. For our study, participants will be scored from 1-6 on this scale, with scores of 1-2 indicating no frailty, 4-5 indicating pre-frailty and 6 indicating frailty. Therefore, higher scores will indicate a worse outcome regarding frailty severity.
Electronic Frailty Index | Initial patient screening (within clinic of Nottingham University Hospitals)
  The Electronic Frailty Index will provide information on patient's frailty status already evident in their medical records.
Nottingham Extended Activities of Daily Living Scale | Baseline (During visit to University physiology laboratory)
  This questionnaire assesses participant's independence in daily tasks (e.g. housework, feeding). Participants will be scored from 0-22, with higher scores indicating greater independence when performing daily activities.
Fried frailty phenotype | Baseline (During visit to University physiology laboratory)
  Participant's score on the frailty phenotype will be assessed by two functional measures (walking speed and hand grip strength) and three self report measures (questionnaires assessing exhaustion, physical activity levels and weight loss).
Minnesota Leisure Time Activity Questionnaire | Baseline (During visit to University physiology laboratory)
  Participant's duration and type of physical activity will be assessed using a modified version of the Minnesota Leisure Time Activity Questionnaire, as part of the Fried frailty phenotype assessment.
Center for Epidemiologic Studies Depression Scale | Baseline (During visit to University physiology laboratory)
  Participant exhaustion will be determined using the Center for Epidemiologic Studies Depression Scale, as part of the Fried frailty phenotype assessment. Participants will be scored from 0-60, with higher scores indicating the presence of more depressive symptoms.
Montreal Cognitive Assessment questionnaire | Baseline (During visit to University physiology laboratory)
  The cognitive function of participants will be assessed using the Montreal Cognitive Assessment questionnaire.
Knee extension power output | Baseline (During visit to University physiology laboratory)
  Power output of the quadriceps muscles will be assessed using a Cybex dynamometer, during separate sets of slow and fast isokinetic contractions.
Knee extension fatigability | Baseline (During visit to University physiology laboratory)
  Fatigability of the quadriceps muscles will be assessed using a Cybex dynamometer, during separate sets of slow and fast isokinetic contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Taylor, PhD student, Principal Investigator — University of Nottingham; Tahir Masud, Professor, Principal Investigator — Nottingham University Hospitals NHS Trust; Paul Greenhaff, Professor, Principal Investigator — University of Nottingham; Susan Francis, Professor, Principal Investigator — University of Nottingham; John Gladman, Professor, Study Chair — University of Nottingham
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Fried LP, Xue QL, Cappola AR, Ferrucci L, Chaves P, Varadhan R, Guralnik JM, Leng SX, Semba RD, Walston JD, Blaum CS, Bandeen-Roche K. Nonlinear multisystem physiological dysregulation associated with frailty in older women: implications for etiology and treatment. J Gerontol A Biol Sci Med Sci. 2009 Oct;64(10):1049-57. doi: 10.1093/gerona/glp076. Epub 2009 Jun 30. PMID 19567825